CLINICAL TRIAL: NCT03801564
Title: Efficacy of Intra-articular Injections of Hyaluronic Acid and Platelet-rich Plasma for Patients With Knee Osteoarthritis: Changes in Function, Quality of Life and Cartilage Loss as Assessed by Magnetic Resonance Imaging
Brief Title: Knee Osteoarthritis: Platelet Rich Plasma or Hyaluronic Acid
Acronym: OA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Antalya Training and Research Hospital (Other Government)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Naciye Fusun Toraman, Professor, Antalya Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 118S014
Record Dates: First submitted 2019-01-04; First posted 2019-01-11 (Actual); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Knee Osteoarthritis
Keywords: Knee Osteoarthritis; Hyaluronic Acid; Platelet Rich Plasma
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: The volunteer, sedanter patients with Kellgren Lawrence (KL) radiological grade II-III knee OA, unilateral knee pain, aged 50-70 years will be selected. Exclusion criterias are; KL radiological grade ≥2 of contrlateral knee, thrombocytopenia, coagulopathy, OA of multiple joints, acute exacerbation of any joint, intraarticular steroid, PRP or HA injection within 6 months, non-steroidal anti inflammatory drugs or steroid use within 6 weeks; diabetes and cancer; severe anemia (Hb <10), presence of heart and lung disease that can not perform physical function tests, secondary inflammatory arthritis; knee surgery or knee injury; planning for joint replacement within the next 3 months, difficulty in answering the questionnaires, limitation in joint range of motion, presence of genu varum/valgum >50. Patients will be divided into two groups: Group 1: HA group, Group 2: PRP group, using covariate adaptive randomization as age and osteoarthritis severity covariate.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: There are five investigators in this study. N.Fusun Toraman is project manager and blind for the study groups. Yasemin Karaman and Sevim Yıldız are radiologists and blind for the study groups. Meral Bilgilisoy Filiz and Aslı Karadag Ozdemir know the groups, they will select the participants, and Meral Bilgilisoy Filiz will apply intraarticular injections via ultrasound. The participants of the groups do not know each other.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Platelet Rich Plasma Group (PRP) (Experimental): Platelet Rich Plasma Treatment Group (PRP): The blood is drawn from the antecubital vein to the 10cc line of EasyPRP syringe consisted 1.5ml of anticoagulant. The syringe is centrifuged at a rate of 1200 g for 2 minutes. Then the syringe is rotated and the lower chamber filled with erythrocytes is discharged. The connector is inverted and the air gap is discharged. The injector is again centrifuged at 1200G for 10 minutes. Then the injector is rotated in the direction of the arrow, the lower stopper is removed. The application injector of 3cc with connector is placed in the EasyPRP injector. 1 ml of the PRP containing Buffycoat is separated for content analysis, the remaining 2 ml of the string is injected. Injection is repeated one month interval
  Interventions: Device: Platelet Rich Plasma Treatment Group (PRP)
- Hyaluronic acid Group (HA) (Experimental): Hyaluronic Acid Treatment Group (HA): 2 ml HA (32mg / ml) containing 1.6% sodium hyaluronate is injected intraarticular. The molecular weight is 800 - 1200 K Dalton. The viscosity is 20 pascal / s. The pH of the product is 7-7.5.Injection is repeated one month interval.
  Interventions: Device: Hyaluronic Acid Treatment Group (HA)

INTERVENTIONS:
Device: Platelet Rich Plasma Treatment Group (PRP) — EASY PRP is in category IIa and manufactured by Neotec Biotechnology Industry and Foreign Trade Company. (Item No. 8680976403603; UNSPSC 42295470; GMDN 46923; certificate no: M.2016.106.7294).
  Arms: Platelet Rich Plasma Group (PRP)
Device: Hyaluronic Acid Treatment Group (HA) — REGENFLEX STARTER is a class III intraarticular viscosupplementation device (Art. No. 8681065100076; UNSPSC 42295509). Sodium hyaluronate is obtained by bacterial fermentation (STREPTOCOCCUS EQUI) method. The product is in disposable packages, sterile and contained in a 2 ml pyrogen-free syringe.
  Arms: Hyaluronic acid Group (HA)

SUMMARY:
PURPOSE: To compare the effect of hyaluronic acid (HA) or platelet-rich plasma (PRP) on pain, physical function, quality of life and knee joint morphology in patients with knee osteoarthritis severity II-III.

BACKGROUND: Knee osteoarthritis affects quality of life significantly because it is the most common joint disease and causes considerable disability. Pathogenesis is multifactorial, nevertheless reduced cartilage production, increased destruction, and synovial inflammation are important factors in the osteoarthritis process. Today, symptomatic drugs are commonly used in the treatment of osteoarthritis, but these treatments have limited effects on cartilage degeneration. Intraarticularly, hyaluronic acid (HA) and platelet-rich plasma (PRP) treatments have been used for osteoarthritis due to pain and functional effects. HA has been shown to reduce the levels of collagen degradation products and maintain normal cartilage metabolism. PRP is thought to have positive effects on clinical and tissue healing due to the numerous growth factors involved. However there is no research to prove definitively that one of the two applications in knee osteoarthritis is superior to the other.

METHOD: 120 patients between the ages of 50-70, OA severity II-III will be included in the study. Patients will be stratified according to the severity and age of OA, and two groups will be randomly assigned as HA and PRP. HA and PRP injections will be performed two times and one month apart. Outcome measures are pain, physical function, quality of life, muscle strength, WORMS, and patient satisfaction. Each patient will be examined at baseline, first, third, sixth, ninth and twelfth months.

DETAILED DESCRIPTION:
PROJECT TEAM N.Fusun Toraman (NFT) cell phone: +90 505 355 9045 e.mail: fusuntoraman@gmail.com Meral Bilgilisoy Filiz (MBF) cell phone: +90 505 647 5840 e.mail: mbilgilisoy@gmail.com Aslı Karadag Ozdemir (AKO) cell phone: +90 555 276 6334 e.mail:aslikaradagoz@gmail.com Yasemin Karaman (YK) cell phone: +90 533 375 0070 e.mail: dryaseminkaraman@hotmail.com Sevim Yıldız (SY) cell phone: +90 535 967 3870 e.mail: syildiz07@yahoo.com

PROJECT PRESENTATION AND ETHICAL APPROVAL The project team and the physicians of the Physical Therapy and Rehabilitation Clinic were informed about the research topic, content and applications and their suggestions were recorded (August 2017). The research was submitted to the Antalya Training and Research Hospital Ethical Committee and Ethic approval was obtained (September 21, 2017 / Decision number 2017-177). The research was presented as a 3001-TUBITAK project on December 2017, and Contract is signed (September 07, 2018 / Project number 118S014). Project start date was determined as September 21, 2018 by TUBITAK.

The Contract of Project was submitted to the Research and Development Office of Antalya Training and Research Hospital and Purchasing Officers were determined by them (September 13, 2018 / 00076415138). Technical specifications were prepared for the purchase of Regenflex Starter and EasyPRP, bidding process was made, contract was written and products purchased (October 30, 2018 / 00079677083). Technical specification was prepared for the purchase of the computer, bidding process was made, contract was prepared and computer purchased (October 02, 2018 / 00077859953). Technical specification was prepared for the laboratory testing, bidding process was made, contract was prepared (November 22, 2018).It was learned that the research project should be sent to Turkey Pharmaceuticals and Medical Devices Agency Department of Clinical Research at the meeting entitled as Good Clinical Researches which was held on November 30, 2018, at Ministry of Health, Ankara. The project was sent to Turkey Pharmaceuticals and Medical Devices Agency Department of Clinical Research on December 17, 2018 and start time of the project was changed to January 07, 2019. The mandatory amendment on the commencement date of the project was reported to TUBITAK by writing an official letter with attached information related with the Basic Principles of Clinical Trials. Additionally, a similar official letter sent to TUBITAK was written to the Ethical Committee of Antalya Training and Research Hospital and Clinical Research and Development Unit on December 19, 2018.The project is approved by Turkey Pharmaceuticals and Medical Devices Agency Department of Clinical Research (January 03, 2019/No:71146310-511.06-E.1116/subject:2018-157) PATIENT RECRUITMENT: Hospital records of patients admitted to Outpatient Clinics of Physical Therapy and Rehabilitation with the diagnostic code M17.0-M17.9, M24.1, M25.5, between 50-79 ages, and between March and August 2018 were controlled in order to determine how many months were necessary for patient selection and radiological results of the patients were evaluated. At the end of the evaluation, it was decided that two months of the patient recruitment time were sufficient. It is decided to recruit the patients diagnosed as knee osteoarthritis after clinical, laboratory and radiological examination and referred to the project team between January and March 2019. Diagnosis of the knee osteoarthritis is made according to American College of Rheumatology diagnostic criterias. The patients are informed about the content of the study by the principal investigator and the research assistant (NFT, and AKO, respectively]. The criterias of inclusion and exclusion, follow-up times and importance of follow-up are explained to the patients and consent is obtained from the patients who meet the criteria. NFT ve AKO examine the patients and select the patients using inclusion and exclusion criterias. If the sufficient number of patients do not meet the criterias for inclusion between the dates specified, the patients are referred from Physical Therapy and Rehabilitation Outpatient Clinics of Ataturk State Hospital. The patients are selected using the inclusion and exclusion criterias.

ASSESSMENT PROCEDURE: NFT and AKO get information related with age, sex, medical and family history, comorbidities, menopausal characteristics of the female patients, radiologic and laboratory diagnostic tests, education, occupation, socioeconomic status, habits, medication use, cognitive level, physical activity status, dominant extremity. Then activity and rest pain is asked, body composition, physical performance tests, and isokinetic test are applied, questionnaires of disease-specific and overall quality of life are filled. Under AKO supervision physical performance tests are performed by a single occupational therapist, and isokinetic test and body composition measures are performed by a single physiotherapist. The weight-bearing knee radiologies are evaluated independently by SY and NFT according to Kellgren Lawrence criterias. Randomization is performed by MBF after all examinations are completed. The groups are stratified as PRP and HA using covariate adaptive randomization as age and osteoarthritis severity covariate.MRI is performed after appointment of radiology department. Two of MRI in the morning and two of MRI in the afternoon are performed daily. The patients who can not perform MRI examinations are recommended to undergo sedation. The patients who do not want to undergo MRI with sedation are excluded from the study by establishing the definition of non-volunteers. MRI is performed at the beginning and at the end of the study and the evaluation will be made by the two radiologist independently (SY, and YK). Total of 16 patients- eight patients of the HA group in the morning time, eight of the patients of the PRP group in the afternoon as daily- are injected by MBF. Injections are performed by using suprapatellar intraarticular route, ultrasound guided and 20G injector and are repeated after one month. Three passive flexion and extension movement is performed after injection, and after fifteen minutes of the rest the patient is sent to home. On the day of the injection, it is recommended that the patient does not perform intensive activities for 24 hours and should not remain standing for a long time. If there is pain and swelling on the knee, it is recommended to use 500 mg of paracetamol which does not contain codeine, cold application three times a day and not to use nonsteroid antiinflammatory medicines. If pain persists, it is recommended to communicate with the physiatrist who performs injection (MBF).Exercise brochure is prepared for both of the groups to be performed one day after injection and is recommended to continue for one year. Cold application, analgesic and NSAID use, exercise compliance/adherence, and adverse events related with the injections are asked to the patients on each of the evaluation time and the results are recorded.Patient satisfaction with a 6-point Likert scale is evaluated on each time of the evaluation. Each of the patient is examined at baseline, and also at the first, at the third, at the sixth, at the ninth and at the twelfth months for all of the outcome measures. MRI is assessed at baseline and at the twelfth month. Follow-up is provided by phone calling and inviting the patient.

DATA COLLECTION PROCEDURE: The groups are encoded and randomized by MBF. The questionnaires are filled by AKO. All of the results of examination, laboratory, radiography and outcome measures will be saved in a separate file for each of the patient by AKO. The data in the files is recorded to the computer by AKO in every weekend. The written files and computer data are checked by MBF.

DATA ANALYSIS PROCEDURE: Dependent variables are pain, physical performance measures, muscle strength, quality of life, patient satisfaction, Whole-Organ Magnetic Resonance Imaging Score (WORMS). Independent variables are PRP and HA. Sample size is determined as a minimum clinical important difference (MCID) of 1.33 on a scale of 0-10 on the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC). It is calculated that at least 46 patients should be in each group as a total sample size of 92 with 0.80 power and a standard deviation of 2.25 by taking into account the MCID in WOMAC. Considering the drop outs, it is decided to take 60 patients for each group and 120 patients in total. Statistical analysis is performed using SPSS version 18. The frequency analysis is used for the demographic data, and the variance homogenity and distribution of the variables are analysed with Levene test and Kolmogorov Smirnov test respectively. The mean and standard deviation are calculated for the baseline outcome measures which are normally distributed and homogen and independent t-test is used to compare the groups. Median, minimum and maximum values are calculated for the baseline outcome measures which are not normally distributed and non-homogen and Mann-Whitney U test is used for the group comparison. The significance is set as p<0.05. The effect of time and group is analysed by using repeated two-way analysis of variance (RM-ANOVA) or two-way analysis of covariance (RM ANCOVA) taking into account the difference in baseline measurements. In RM-ANOVA or RM-ANCOVA tests, the selection of univariate or multivariate approach is selected according to the data distribution, the sphericity and epsilon value. A multivariate approach is chosen for variables which are not normally distributed. The univariate approach is used when the sphericity test is not significant in variables that fulfill the normal distribution assumption. When the sphericity test is significant, the cut-point of epsilon value which is 0.750 is checked. If the epsilon is ≥ 0.750, the highest value of univariate test approach and if the epsilon <0.750 the multivariate approach is recorded. The effect sizes calculated are recorded for group and time effects for RM-ANOVA and RM-ANCOVA tests. The effect sizes are interpreted as follows: negligible effect of between 0.00-0.10, the small effect of between 0.10-0.30, the medium effect of between 0.30-0.50; high effect of between 0.50-0.70; very high effect of between 0.70-0.90, and perfect effect of between 0.90-1.00. The post hoc Bonferroni test is used to compare the group effect and time effect. Significance value for the pain, the quality of life, the muscle strength, the physical function measures, and the patient satisfaction is p <0.01 (0.05/5), and for MRI measure is p <0.025 (0.05/2). MRI results by the two independent researcher (YK and SY) and baseline knee radiology are evaluated by the two independent researcher (SY and NFT). Interobserver reliability for MRI and baseline knee radiology results is calculated by using Pearson or Spearman correlation according to the distribution properties of the variables. The correlation between pain, physical function, muscle strength and magnetic resonance change will be calculated by Pearson or Spearman correlation according to the variables distribution properties. Mean imputation technique is used for missing values on a variable. All of the statistical analysis is performed by NFT and is checked by Full Software Engineering Advertising Promotion Tourism Organization Industry Trade Limited Company.

ELIGIBILITY:
Inclusion Criteria:

* Between 50-70 years of age
* Kellgren Lawrence (KL) radiological grade II-III knee OA
* Sedanter
* Unilateral knee pain
* Volunteer

Exclusion Criteria:

* KL radiological grade ≥2 of contrlateral knee
* Thrombocytopenia (<150.000/mm3)
* Coagulopathy
* Osteoarthritis of multiple joints
* Acute exacerbation of any joint
* Intraarticular steroid, PRP or HA injection within 6 months
* Non-steroidal anti inflammatory drugs or steroid use within 6 weeks
* Diabetes and cancer
* Severe anemia (hemoglobin <10)
* Presence of heart and lung disease that can not perform physical function tests
* Secondary inflammatory arthritis
* Knee surgery or knee injury
* Planning for joint replacement within the next 3 months
* Difficulty in answering the questionnaires
* Limitation in joint range of motion
* Presence of genu varum / valgum >50.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-01-07 (Actual); Primary Completion 2020-01-07 (Estimated); Study Completion 2020-03-07 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Health Related Quality of Life Measured by Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Periodically During 12 Months | The scale is filled before the first and second injection which is one month apart, then the evaluation continues at 3rd, 6th, 9th, and 12th month.
  The validated and reliable Turkish version of WOMAC consisted of three subscales- pain, stiffness, and physical function. Subscale of pain score range is between 0-20; stiffness score range is between 0-8; physical function score range is between 0-68. Values are summed up and the correction factors are used which are 0.50 for pain, 1.25 for stiffness, 0.147 for physical function to obtain total score. Total WOMAC score is between 0-100 and the higher scores indicate the greater disease severity.

SECONDARY OUTCOMES:
Change from Baseline Pain measured by Visual Analogue Scale (VAS) Periodically During 12 Months | VAS is evaluated before the first and second injection which is applied one month apart, then the evaluation continues at 3rd, 6th, 9th, and 12th month.
  Activity and rest pain is evaluated on a straight line of fixed length, 100 mm (0 = no pain, 100 = the most severe pain). (Creamer et al., 1999)
Change from Baseline Functional Strength Measured by Chair Stand Test Periodically During 12 Months | The test is evaluated before the first and second injection which is applied one month apart, then the evaluation continues at 3rd, 6th, 9th, and 12th month.
  The patient stands up completely up from the sitting position, then completely backs down. The score is the total number of stands executed correctly within 30 seconds. The time in seconds is recorded using stop-watch (McAlindon et al., 2015).
Change from Baseline Strength and Balance Measured by Stair Ascend/Descend Test Periodically During 12 months | The test is evaluated before the first and second injection which is applied one month apart, then the evaluation continues at 3rd, 6th, 9th, and 12th month.
  The patient ascends and descends a flight of stairs (10-step stair) separately as soon as possible without handrail. The time in seconds is recorded using stop-watch (McAlindon et al., 2015).
Change from Baseline Agility Measured by Timed Up-and-Go (TUG) Test Periodically During 12 months | The test is evaluated before the first and second injection which is applied one month apart, then the evaluation continues at 3rd, 6th, 9th, and 12th month.
  The patient sitting in the chair, gets up, walks 3 meters without aid, walks back to the chair, then sits down. The score is the shortest time to rise from a chair, and return to the seated position. The time in seconds is recorded using stop-watch (McAlindon et al., 2015).
Change from Baseline Endurance Measured by 6 Min Walk Test Periodically During 12 Months | The test is evaluated before the first and second injection which is applied one month apart, then the evaluation continues at 3rd, 6th, 9th, and 12th month
  The patient is asked to walk as fast and as possible in six minutes, between the two cones placed at a distance of 25 meters. The patient may be allowed to stop and then walk within the test period. Time of stop is recorded. The time in seconds is recorded using stop-watch (McAlindon et al., 2015).
Change from Baseline Absolute Strength of Knee Extensor and Flexor Muscle by Isokinetic Test Periodically During 12 Months | The test is evaluated before the first and second injection which is applied one month apart, then the evaluation continues at 3rd, 6th, 9th, and 12th month.
  Test measures absolute muscle strength of the quadriceps and hamstring muscles and is applied in concentric modality in speed of 60 degrees per second (5 repetitions) and 180 degrees per second (10 repetitions) in knee flexion and extension at 10-90 degrees of range of movement with gravity correction for both of the extremities. Absolute peak torque is recorded as Newtonmeter (Nm).
Change from Baseline Relative Strength of Knee Extensor and Flexor Muscle by Isokinetic Test Periodically During 12 Months | The test is evaluated before the first and second injection which is applied one month apart, then the evaluation continues at 3rd, 6th, 9th, and 12th month.
  Test measures relative strength of the quadriceps and hamstring muscles and is applied in concentric modality in speed of 60 degrees per second (5 repetitions) and 180 degrees per second (10 repetitions) in knee flexion and extension at 10-90 degrees of range of movement with gravity correction for both of the extremities. Relative peak torque is recorded as peak torque-to body weight ratio (Nm/kg)
Change from Baseline Average Power of Knee Extensor and Flexor Muscle by Isokinetic Test Periodically During 12 months | The test is evaluated before the first and second injection which is applied one month apart, then the evaluation continues at 3rd, 6th, 9th, and 12th month.
  Test measures average power of the quadriceps and hamstring muscles and is applied in concentric modality in speed of 60 degrees per second (5 repetitions) and 180 degrees per second (10 repetitions) in knee flexion and extension at 10-90 degrees of range of movement with gravity correction for both of the extremities. Muscular average power is recorded as Watt (W).
Change from Baseline Health Status Measured by Nottingham Health Profile (NHP) Periodically During 12 Months | The scale is evaluated before the first and second injection which is applied one month apart, then the evaluation continues at 3rd, 6th, 9th, and 12th month.
  NHP is a scale developed to measure perceived health. Turkish version of the scale used consists of two parts (Kucukdeveci et al, 2000). Part I contains 38 yes/no items that assess 6 subscales (pain, physical mobility, emotional reactions, energy, social isolation and sleep). The each question answered by yes is assigned a weighted value. Scores for each subscale can range from 0 to 100. Total score range of NHP is between 0-600. Part II contains 7 general yes/no questions concerning daily living problems and score range is between 0-7, with a higher score indicating greater distress for Part I and II.
Change from Baseline Whole Organ MRI Scoring Periodically During 12 Months | The test is evaluated before the first and second injection which is applied one month apart, then the evaluation continues at 3rd, 6th, 9th, and 12th month.
  Magnetic Resonance Images are scored with respect to 14 independent features of patellofemoral joint (PFJ),medial femorotibial joint(MFTJ), lateral femorotibial joint (LFTJ), and non-articulating portion of the tibial plateau (S). Total cartilage score range is between 0-84; total marrow abnormality and bone cysts range are between 0-45; total bone attrition range is between 0-42; total osteophyte range is between 0-98; total compartment range is 0-35 for MFTJ, LFTJ, and 0-28 for PFJ; total menisci score range is between 0-12,ligaments score range is between 0-12, synovitis score range is between 0-3. Subscales are summed for the total WORMS score whic is between 0-332 and the higher values represent a worse outcome.Additionally tendon abnormalities, avascular necrosis,stress fracture,insufficiency fracture,osteochondral fracture,tumors, and technical limitations that interfered with the reliability of the scoring are specified and noted. (Peterfy et al, 2004).
Change from Patient Satisfaction Related with Treatment Periodically During 12 Months | Patient satisfaction is evaluated before the first and second injection which is applied one month apart, then the evaluation continues at 3rd, 6th, 9th, and 12th month.
  The patient's global satisfaction related with the treatment is evaluated with a 6-point scale showing that the patient extremely satisfied from the treatment (1 point) and the patient extremely dissatisfied from the treatment (6 point) (Hoeksma et al, 2006).
Change from Baseline Body Weight (BW) Periodically During 12 Months | BW is evaluated before the first and second injection which is applied one month apart, then the evaluation continues at 3rd, 6th, 9th, and 12th month.
  BW is evaluated using TANITA MC-180MA and is recorded as kg.
Change from Baseline % Fat Periodically During 12 Months | % fat is evaluated before the first and second injection which is applied one month apart, then the evaluation continues at 3rd, 6th, 9th, and 12th month.
  % fat is evaluated using TANITA MC-180MA and is recorded as percentile value.
Change from Baseline Body Mass Index (BMI) Periodically During 12 Months | BMI is evaluated before the first and second injection which is applied one month apart, then the evaluation continues at 3rd, 6th, 9th, and 12th month.
  BMI is evaluated using TANITA MC-180MA and is recorded kg/square meter.

CONTACTS AND LOCATIONS:
Overall Officials: NFusun Toraman, Prof, Principal Investigator — Ministry of Health Antalya Training and Research Hospital; Meral Bilgilisoy Filiz, MD,PM&R, Study Chair — Ministry of Health Antalya Training and Research Hospital; Yasemin Karaman, MD,Radiology, Study Chair — Ministry of Health Antalya Training and Research Hospital; Sevim Yildiz, MD,Radiology, Study Chair — Ministry of Health Sancaktepe Training and Research Hospital; Asli Karadag Ozdemir, MD,Res.Ass., Study Chair — Health Sciences University Antalya Training and Research Hospital
Locations (1):
- Naciye Fusun Toraman, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Creamer P, Lethbridge-Cejku M, Hochberg MC. Determinants of pain severity in knee osteoarthritis: effect of demographic and psychosocial variables using 3 pain measures. J Rheumatol. 1999 Aug;26(8):1785-92. PMID 10451078
- [Background] McAlindon TE, Driban JB, Henrotin Y, Hunter DJ, Jiang GL, Skou ST, Wang S, Schnitzer T. OARSI Clinical Trials Recommendations: Design, conduct, and reporting of clinical trials for knee osteoarthritis. Osteoarthritis Cartilage. 2015 May;23(5):747-60. doi: 10.1016/j.joca.2015.03.005. PMID 25952346
- [Background] Tuzun EH, Eker L, Aytar A, Daskapan A, Bayramoglu M. Acceptability, reliability, validity and responsiveness of the Turkish version of WOMAC osteoarthritis index. Osteoarthritis Cartilage. 2005 Jan;13(1):28-33. doi: 10.1016/j.joca.2004.10.010. PMID 15639634
- [Background] Kucukdeveci AA, McKenna SP, Kutlay S, Gursel Y, Whalley D, Arasil T. The development and psychometric assessment of the Turkish version of the Nottingham Health Profile. Int J Rehabil Res. 2000 Mar;23(1):31-8. doi: 10.1097/00004356-200023010-00004. PMID 10826123
- [Background] Peterfy CG, Guermazi A, Zaim S, Tirman PF, Miaux Y, White D, Kothari M, Lu Y, Fye K, Zhao S, Genant HK. Whole-Organ Magnetic Resonance Imaging Score (WORMS) of the knee in osteoarthritis. Osteoarthritis Cartilage. 2004 Mar;12(3):177-90. doi: 10.1016/j.joca.2003.11.003. PMID 14972335
- [Background] Hoeksma HL, van den Ende CH, Breedveld FC, Ronday HK, Dekker J. A comparison of the OARSI response criteria with patient's global assessment in patients with osteoarthritis of the hip treated with a non-pharmacological intervention. Osteoarthritis Cartilage. 2006 Jan;14(1):77-81. doi: 10.1016/j.joca.2005.07.019. Epub 2005 Oct 7. PMID 16214379